CLINICAL TRIAL: NCT04580771
Title: IMMUNOCERV: Evaluating the Safety of Chemoradiation Combined With PDS0101 Immunotherapy in Treating Locally Advanced Cervical Cancer
Brief Title: A Vaccine (PDS0101) and Chemoradiation for the Treatment of Stage IB3-IVA Cervical Cancer, the IMMUNOCERV Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1260; NCI-2020-06810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1260 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB3 Cervical Cancer FIGO 2018; Stage II Cervical Cancer FIGO 2018; Stage IIA Cervical Cancer FIGO 2018; Stage IIA1 Cervical Cancer FIGO 2018; Stage IIA2 Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018; Stage III Cervical Cancer FIGO 2018; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IIIC Cervical Cancer FIGO 2018; Stage IIIC1 Cervical Cancer FIGO 2018; Stage IIIC2 Cervical Cancer FIGO 2018; Stage IVA Cervical Cancer FIGO 2018
MeSH Terms: interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, cisplatin, PDS0101) (Experimental): Patients undergo radiation therapy over 1 hour 5 days per week (Monday-Friday) for 5-7 weeks and receive cisplatin IV over 4 hours QW during the 5 weeks of radiation therapy in the absence of disease progression and unacceptable toxicity. Patients also receive PDS0101 SC on days -10, 7, 28, 49, and 170 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Biological: Liposomal HPV-16 E6/E7 Multipeptide Vaccine PDS0101; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Biological: Liposomal HPV-16 E6/E7 Multipeptide Vaccine PDS0101 — Given SC
  Other Names: mmunoMAPK-RDOTAP /HPV-16 E6/E7 Peptide Antigen Vaccine; PDS0101
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase IIA trial studies the effect of a vaccine (PDS0101) when given together with chemotherapy and radiation therapy (chemoradiation) in treating patients with stage IB3-IVA cervical cancer. Chemotherapy drugs, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. PDS0101 is a type of vaccine that is intended to help the immune system respond to human papillomavirus (HPV16)-infected cervical tumor cells. PDS0101 contains two active components: the first is called R-DOTAP (Versamune) and is included in the vaccine to boost the immune system's response against the HPV viral proteins and the second group of active components are selected small pieces of proteins (called peptides) taken from the HPV virus. Giving PDS0101 in combination with chemoradiation may work help to control cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and toxicity profile of delivering the immune nanoparticle liposomal HPV-16 E6/E7 multipeptide vaccine PDS0101 (PDS0101) with standard-of-care chemoradiation (chemoRT) in patients with locally advanced cervical cancer.

SECONDARY OBJECTIVES:

I. Rate of complete metabolic response on day 170 (+/- 14 days) positron emission tomography computed tomography (PET CT).

II. Rate of >= 90% gross tumor volume reduction day 35 magnetic resonance imaging (MRI) (+/- 5 days).

III. Report rates of local control (LC), progression-free survival (PFS), and overall survival (OS) at 12 and 18 months following chemoRT completion.

IV. Long-term safety: rate of grade >= 3 chronic toxicity (from day 81 to completion of trial).

EXPLORATORY HPV-SPECIFIC IMMUNE RESPONSE OBJECTIVES:

I. Enzyme-linked immunosorbent spot (ELISpot) assays on interferon-gamma and granzyme B levels in E6/7-specific T cells isolated from peripheral blood mononuclear cells (PBMCs).

II. Compare intratumoral T-cell receptor (TCR) clonality at baseline and end of treatment by TCR sequencing.

III. Measure CD4+ and CD8+ tumor-infiltrating lymphocytes (TILs) from cervical brush samples by using markers of T-cell exhaustion (PD1, CTLA4) and T cell-activation (granzyme B, CD69+).

IV. Assess the intestinal and cervical microbiome by analyzing rectal and cervical swab samples with 16s ribosomal ribonucleic acid (rRNA) sequencing.

V. Additional assays such as circulating tumor cells, circulating cell-free tumor deoxyribonucleic acid (DNA) (ccfDNA), and other assays will be performed at the discretion of the principal investigator.

OUTLINE:

Patients undergo radiation therapy over 1 hour 5 days per week (Monday-Friday) for 5-7 weeks and receive cisplatin intravenously (IV) over 4 hours once per week (QW) during the 5 weeks of radiation therapy in the absence of disease progression and unacceptable toxicity. Patients also receive PDS0101 subcutaneously (SC) on days -10, 7, 28, 49, and 170 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 1, 4, 6, 12, and 18 weeks, and 18 months.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older
2. Newly diagnosed locally advanced squamous cell carcinoma of cervix (FIGO 2018 stage IB3-IVA with primary tumor ≥ 5 cm and/or positive pelvic or periaortic nodal disease assessed by imaging).
3. Histologic diagnosis of squamous cell carcinoma of the cervix.
4. Written informed consent before initiation of any study-related procedures;
5. WHO/ECOG performance status 0-2.
6. Adequate liver (ALT, AST, Alk Phos and total Bili ≤ 2-fold the upper limit of normal), and renal functions (Creatinine ≤ 1.5).
7. Absence of current malignancies at other sites, except for adequately treated basal or squamous cell carcinoma of the skin. Cancer survivors who have undergone potentially curative therapy for a prior malignancy who have no evidence of that disease for 5 years and who are deemed at low risk for recurrence are eligible for the study

Exclusion Criteria:

1. HIV infection, cellular immune deficiencies, hypogammaglobulinemia or dysgammaglobulinemia, or hereditary or congenital immunodeficiencies
2. Prior diagnosis of hepatitis B or C (unless anti-hepatitis C therapy has produced a sustained virologic response);
3. History of clinically significant autoimmune disease, Crohn's disease, or ulcerative colitis
4. Serious concomitant disorder, including active systemic infection requiring treatment, as judged by the Investigator.
5. Receipt of immunotherapy (e.g., IFNs, check-point inhibitors, tumor necrosis factor, interleukins, etc.) or biological response modifiers (GM-CSF, granulocyte colony-stimulating factor, macrophage colony-stimulating factor) within 4 weeks before the first study vaccination.
6. Receipt of chronic systemic steroid therapy (in dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

   • Current or recent use of physiologic doses of intra-articular, topical, or inhaled corticosteroids is acceptable.
7. History of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines [e.g., Silgard®, Cervarix®, Gardasil®] are not excluded)
8. Known or suspected hypersensitivity to any component of the investigational product or contraindications to cisplatin (e.g., peripheral neuropathy grade ≤ 2 or ototoxicity ≤grade 2 per CTCAE v5.0)
9. Previous pelvic RT.
10. Previous chemotherapy for the cervix tumor
11. Previous hysterectomy or will have a hysterectomy as part of their initial cervical cancer therapy
12. Prior major surgery within 4 weeks of enrollment from which the patient has not recovered
13. Other condition or prior therapy that, in the opinion of the Investigator, compromises the subject's welfare or may confound study results
14. Concurrent participation in another therapeutic investigational study or use of another investigational drug within 6 months before the first study vaccination
15. Previous enrollment in this study
16. HPV genotyping is to be done from cervical swab samples. Enrollment will not require HPV testing.
17. Pregnancy: a female subject defined as a WOCBP who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
Rate of grade >= 3 acute toxicity | Day -10 to day 80
  Measured from first vaccine injection up to 30 days following completion of chemoradiotherapy (chemoRT). Adverse events (AEs) will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Any AE that occurs between the first day of PDS0101 injection and up to 30 days following completion of chemoRT (~Day 80) will be considered as acute toxicity (AT).

SECONDARY OUTCOMES:
Rate of complete metabolic response | Day 170
  Measured by positron emission tomography computed tomography (PET CT).
Rate of >= 90% gross tumor volume reduction | Day 35
  Measured by magnetic resonance imaging (MRI).
Rates of local control | At 12 and 18 months
  Will be represented by Kaplan-Meier curves.
Rates of progression-free survival | At 12 and 18 months
  Will be represented by Kaplan-Meier curves.
Rates of overall survival | At 12 and 18 months
  Will be represented by Kaplan-Meier curves.
Rate of grade >= 3 chronic toxicity | Day 81 to completion of trial
  AEs will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Chronic toxicity (CT) is any toxicity that occurs outside of the AT window (between Days 81 and study completion of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Klopp, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org